CLINICAL TRIAL: NCT01173757
Title: A Phase I, Healthy Volunteer Determination Of 5HT4 Receptor Occupancy Of PF-04995274, Using PET With Ligand [11C]PF-05127401.
Brief Title: To Evaluate The Relationship Between Plasma Drug Levels And Receptor Binding In Brain Using PET (Positron Emission Tomography) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: B1661002
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04995274 (Experimental)
  Interventions: Drug: PF-04995274

INTERVENTIONS:
Drug: PF-04995274 — Single dose of up to 5 mg PF-04995274, delivered in solution on study day 1

SUMMARY:
The purpose of this study is to evaluate the relationship between plasma drug levels and receptor binding in brain using PET; and to evaluate safety and tolerability after a single administration of PF-04995274 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening
* Fulfillment of any of the MRI contraindications on the standard radiography screening questionnaire

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Exposure response of overall 5HT4 receptor occupancy of PF-04995274 | up to 3 days
5HT4 receptor occupancy by PF-04995274 at regions of interest within the human brain | up to 3 days

SECONDARY OUTCOMES:
Adverse events | up to 3 days
change from baseline in vital signs | up to 3 days
Singlet ECG post-dose | up to 3 days
Clinical safety laboratory endpoints | up to 3 days
Clinical examinations | up to 3 days
Cmax, Tmax, AUClast, and AUCinf for PF-04995274 in plasma | up to 3 days
Cmax, Tmax, AUClast, and AUCinf for PF-05082547 in plasma | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1661002&StudyName=To%20Evaluate%20The%20Relationship%20Between%20Plasma%20Drug%20Levels%20And%20Receptor%20Binding%20In%20Brain%20Using%20PET%20%28Positron%20Emission%20Tomography%29%20In%20He